CLINICAL TRIAL: NCT04879069
Title: Polish Multicenter Pulmonary Embolism Response Teams Outcomes Registry
Brief Title: Polish Multicenter PERTs PE Outcomes Registry
Acronym: PolPERTs
Status: Recruiting | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: Polish Cardiac Society (Other)
Responsible Party: Principal Investigator, Aleksander Araszkiewicz, Professor of Medicine, Poznan University of Medical Sciences
Other Study IDs: 276/21
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Embolism With Acute Cor Pulmonale
Keywords: pulmonary embolism, pulmonary embolism response team,
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intermediate-high risk PE: Confirmed PE causing right ventricle dysfunction confirmed by computed tomography pulmonary angiography or transthoracic echocardiography and elevated troponin level
- High-risk PE: Confirmed PE causing hemodynamic instability:
  1. Cardiac arrest (need for cardiopulmonary resuscitation) or,
  2. Obstructive shock (systolic blood pressure < 90 mmHg or vasopressors required to achieve a systolic blood pressure ≥90 mmHg despite adequate filling status and end-organ hypoperfusion), or
  3. Persistent hypotension (systolic blood pressure < 90 mmHg for at least 15 minutes)

SUMMARY:
Pulmonary embolism (PE) is the third leading cause of cardiovascular mortality. The Pulmonary Embolism Response Team (PERT) concept offers a rapid and multidisciplinary approach focused on improving outcomes for patients with PE. All institutionalized PERTs in Poland have been invited to join the study. The goal of this registry is to describe current practice and outcomes in patients with acute PE treated by Polish PERTs.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is the third leading cause of cardiovascular mortality. The presentation of PE may vary from asymptomatic or mild exertion disturbances (low-risk PE) treated with anticoagulants only to hemodynamic "obstructive" collapse and death (high-risk PE). Patient outcome depends on ability of the right ventricle to sustain the increased afterload caused by the embolic burden. Careful risk stratification is crucial, and the Pulmonary Embolism Response Team (PERT) concept offers a rapid and multidisciplinary approach focused on improving outcomes for patients with PE by advancing its recognition, diagnosis, and treatment. All institutionalized PERTs in Poland have been invited to join the study. The data is administrated by the Poznan University of Medical Sciences on the basis of an agreement between the PERT centres.

The goal of this registry is to describe current practice and outcomes in patients with acute PE guided by Polish PERTs. The primary data recorded include details of each patient's clinical status, co-morbidities, the administered treatment modalities, the results of additional studies (ab tests results, ECG, imaging studies), and the outcome.

The data collection will have no impact on the way the patient is diagnosed and treated.The study endpoints comprise respiratory failure, shock, death distal systemic embolization (i.e. stroke) and major or minor bleeding complications classified according to the International Society on Thrombosis and Haemostasis classification.

ELIGIBILITY:
Inclusion Criteria:

1. PE confirmed by computed tomography pulmonary angiography.
2. PE symptoms duration ≤ 14 days.
3. High-risk PE with hemodynamic instability (one of):

   * cardiac arrest
   * obstructive shock
   * persistent hypotension.
4. Intermediate-high risk PE patients with right ventricle dysfunction confirmed by imaging studies and elevated troponin level.

Exclusion Criteria:

1. Refusal to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients hospitalized due to high-risk or intermediate-high risk PE.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement during hospitalization | 24 hours after specific PE treatment implementation
  Incidence of arterial blood saturation increase >92%
Ventricular strain reduction | 24 hours after specific PE treatment implementation
  Rate of right ventricular strain reduction (right ventricle/left ventricle ratio assessment) in echocardiography
Early mortality rate from pulmonary embolism | Two weeks since PE diagnosis
  Number of patients who died from pulmonary embolism (right heart failure)

SECONDARY OUTCOMES:
Total mortality rate from pulmonary embolism | 3 months since PE diagnosis
  Number of patients who died from pulmonary embolism (right heart failure)
Bleeding events incidence | 3 months since PE diagnosis
  Incidence of major bleedings assessed using ISTH criteria

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Araszkiewicz, Prof., Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, GreaterPoland, Poland

REFERENCES:
- [Derived] Slawek-Szmyt S, Stepniewski J, Kurzyna M, Klaudel J, Kuliczkowski W, Lewandowski M, Grabka M, Roik M, Ordiene R, Jankiewicz S, Kopec G, Darocha S, Mroczek E, Widecka K, Kurzyna P, Lesiak M, Pruszczyk P, Araszkiewicz A. Multicentre, real-world data of next-generation computer-assisted vacuum aspiration thrombectomy in acute pulmonary embolism. Respir Res. 2025 Mar 5;26(1):87. doi: 10.1186/s12931-025-03162-4. PMID 40045310